CLINICAL TRIAL: NCT00289094
Title: Multi-center, Prospective, Clinical Evaluation of the PFC Sigma Rotating Platform Cruciate Retaining Versus PFC Sigma Cruciate Retaining Knee Primary Cases
Brief Title: Randomized Fixed Bearing vs Mobile Bearing Cruciate Retaining TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRP-2
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis; Juvenile Rheumatoid Arthritis; Avascular Necrosis of Bone
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Juvenile; Osteonecrosis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1 (Active Comparator): P.F.C.® Sigma™ Rotating Platform (RP) Cruciate Retaining Knee System
  Interventions: Device: Total Knee Replacement
- 2 (Active Comparator): P.F.C.® Sigma™ Fixed Cruciate Retaining Knee System
  Interventions: Device: Total knee replacement

INTERVENTIONS:
Device: Total Knee Replacement — Rotating Platform (RP) Cruciate Retaining Knee System
  Other Names: P.F.C.® Sigma™ RP Cruciate Retaining Knee System
  Arms: 1
Device: Total knee replacement — Fixed Cruciate Retaining Knee System
  Other Names: P.F.C.® Sigma™ Fixed Cruciate Retaining Knee System
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the rotating platform and fixed bearing implants in patients undergoing primary total knee replacement. Outcome scoring and radiographic assessment will be the methods used to evaluate performance.

DETAILED DESCRIPTION:
This study will evaluate the clinical performance of rotating platform and fixed bearing knee implants. This will be done by obtaining a series of primary total knee replacements. Patients will receive either the P.F.C.® Sigma™ Rotating Platform Cruciate Retaining Knee System or the P.F.C.® Sigma™ Fixed Cruciate Retaining Knee System and assignment is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis
* Rheumatoid Arthritis
* Other inflammatory arthritis
* Avascular necrosis of bone

Exclusion Criteria:

* Prior ipsilateral TKA
* Metabolic disorders
* Joint replacement due to autoimmune disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2001-03-01 (Actual); Primary Completion 2007-12-26 (Actual); Study Completion 2007-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy L O'Dell, EMT, CCRA, CCRC, Study Director — DePuy Orthopaedics
Locations (2):
- United States (2):
  - Billings, Montana
  - Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two US clinical centers performed 99 primary knee replacements in 86 subjects. Recruitment was based on the inclusion and exclusion criteria as specified in the clinical investigation plan.
Pre-assignment Details: Immediately before surgery, the implant type was determined according to the randomization schedule. Before treatment assignment, consented subjects could be excluded from the trial based on results of pre-operative clinical evaluations and/or radiographs, as per the exclusion criteria in the CIP.
Groups:
- Rotating Platform: P.F.C.® Sigma™ Rotating Platform (RP) Cruciate Retaining Knee System has a modular polyethylene insert that is free to rotate around a central pivot point during knee motion.
- Fixed Bearing: P.F.C.® Sigma™ Fixed Cruciate Retaining Knee System implant has a modular polyethylene insert that is intraoperatively locked into position on the metal tibial base.
Period: Overall Study
Arm/Group | Rotating Platform | Fixed Bearing
Started | 50 | 49
Completed | 3 | 2
Not Completed | 47 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotating Platform | Fixed Bearing | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (6.2) | 66.9 (5.1) | 65.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 19 | 23 | 42
Region of Enrollment [Number; unit: participants]
  United States | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Scores
Description: The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. For each section, a score of 80-100 = excellent, 70-79 = good; 60-69 = fair; and < 60 = poor.
Time Frame: Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rotating Platform | Fixed Bearing
Number analyzed (Participants) | 50 | 49
Scores on a scale
  Pre-operative | 40.8 (19.8) | 43.4 (23.0)
  6 months | 84.3 (14.7) | 77.8 (14.9)
  12 months | 86.4 (13.0) | 86.4 (10.0)
  24 months | 89.7 (9.2) | 88.1 (8.8)
  36 months | 92.3 (8.2) | 87.1 (10.4)
  48 months | 94.3 (5.6) | 86.0 (14.7)
  60 months | 95.0 (4.6) | 95.5 (3.5)

2. Secondary Outcome: Complications/Revisions
Time Frame: On-going to end of study.
Reporting Status: Not Posted

3. Secondary Outcome: Medical Imaging
Time Frame: Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.
Reporting Status: Not Posted

4. Secondary Outcome: SF-12 Patient Outcomes
Time Frame: Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Rotating Platform | Fixed Bearing
Serious Adverse Events (participants affected / at risk) | 3/50 | 1/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotating Platform (N=50) | Fixed Bearing (N=49)
Death (General disorders) | 1 (1) | 0 (0)
Femoral Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiacvascular arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less